CLINICAL TRIAL: NCT06759025
Title: Relationship of Kinesiophobia with Clinical Outcomes in Individuals with Chronic Neck Pain
Brief Title: Chronic Neck Pain and Kinesiophobia
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-012
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Chronic Neck Pain
Keywords: chronic neck pain; kinesiophobia; quality of life; functionality
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group

SUMMARY:
In this study, the primary aim was to examine the relationship between kinesiophobia and clinical outcomes in individuals with chronic neck pain. The secondary aim was to compare the level of neck disability, pain, endurance, functionality, muscle and grip strength, and quality of life in individuals with chronic neck pain who had and did not have kinesiophobia; and to determine the determinants of kinesiophobia in patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain complaints that have been ongoing for at least 3 months
* Between the ages of 18-65
* Complaints of numbness and tingling
* Volunteer who can cooperate during communication

Exclusion Criteria:

* History of spinal trauma or surgery
* Neurological, rheumatological, systemic or musculoskeletal problems that affect movement
* Serious comorbidities (such as advanced renal failure, previous history of CVA, malignancy)
* Muscle weakness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusion criteria and are receiving treatment at the Kırşehir Education and Research Hospital Physical Therapy and Rehabilitation Center will constitute the population.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | 24 weeks

SECONDARY OUTCOMES:
Visual Analog Scale | 24 weeks
Neck Disability Index | 24 weeks
Disabilities of the Arm, Shoulder, and Hand Questionnaire | 24 weeks
SF-12 Quality of Life Scale | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No